CLINICAL TRIAL: NCT03777189
Title: Cognitive-Behavioral and Physical Activity Interventions for Binge Eating and Overweight
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: benefits of treatment less than expected
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000023412
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Binge-Eating Disorder; Binge Eating; Overweight and Obesity
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia; Overweight; Obesity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive-Behavioral Therapy (Experimental): Cognitive-behavioral therapy will be delivered in line with recommendations (e.g., NICE 2017). Format will be guided self help with added content related to physical activity.
  Interventions: Behavioral: Cognitive-Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy — Cognitive-behavioral therapy will be delivered in line with recommendations (e.g., NICE 2017). Format will be guided self help with added content related to physical activity.

SUMMARY:
This study aims to perform an open-series pilot trial to examine the efficacy of cognitive-behavioral therapy delivered in a guided self-help format (CBTgsh) with added content related to physical activity (PA), for the treatment of binge-eating disorder (BED), operationalized as BED full diagnostic criteria or BED with the full criteria except for the binge episode size criterion.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years old;
2. Meet DSM-5 criteria for BED or BED but without the size criterion (LOC eating);
3. BMI 25-45 kg/m2;
4. Sedentary activity pattern (< 90 mins/week of moderate-to-vigorous intensity recreational physical activity);
5. Available for the duration of the treatment and follow-up (7 months);
6. Read, comprehend, and write English at a sufficient level to complete study-related materials.

Exclusion criteria:

1. Co-existing psychiatric condition that requires hospitalization or more intensive treatment (e.g., bipolar mood disorders, psychotic illnesses, severe depression).
2. Reports active suicidal or homicidal ideation.
3. Current anorexia or bulimia nervosa.
4. Contraindications to physical activity.
5. Blood pressure >140 systolic or >90 diastolic.
6. Breast-feeding or pregnant, or planning to become pregnant during the study.
7. History of stroke or myocardial infarction.
8. Current or recent (within 12 months) drug or alcohol dependence
9. Currently receiving effective treatment for eating or weight loss.
10. Currently participating in another clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Binge-eating frequency | Post-treatment (4 months)
  Binge eating will be assessed by interview and self-report and the primary outcome is frequency. Frequency will be defined continuously (analyzed dimensionally).
Body mass index | Post-treatment (4 months)
  BMI is calculated using measured height and weight (e.g., percent loss)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Grilo, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States